CLINICAL TRIAL: NCT01865864
Title: Changes In Diurnal Blood Pressure Pattern In Obstructive Sleep Apnea (OSA) Patients After CPAP Therapy
Brief Title: Effect of Continuous Positive Airway Pressure (CPAP) Therapy on Changes of Blood Pressure Between Day and Night
Status: Terminated | Type: Observational
Why Stopped: Difficulty Recruiting subjects
Sponsor: Northwell Health (Other)
Collaborators: Staten Island University Hospital (Other)
Responsible Party: Principal Investigator, Suzanne El-Sayegh, M.D., Northwell Health
Other Study IDs: 07-057
Record Dates: First submitted 2008-12-26; First posted 2013-05-31 (Estimated); Last update posted 2013-05-31 (Estimated); Status verified 2013-05

CONDITIONS: Obstructive Sleep Apnea; Diurnal Blood Pressure
Keywords: CPAP; diurnal blood pressure; obstructive sleep apnea; 24 hour blood pressure monitor
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1: Compliant with CPAP
- 2: noncompliant with CPAP

SUMMARY:
to test whether using CPAP can restore the normal pattern of drop of blood pressure during sleep.

DETAILED DESCRIPTION:
OBJECTIVE:

To investigate the effect of CPAP therapy on the restoration of the normal diurnal blood pressure pattern. Possible improvement of the circadian dipper pattern after CPAP therapy, with or without a decrease in the mean blood pressure, might constitute an additional potential benefit of CPAP therapy in reducing cardiovascular risk in patients with OSA.

STUDY DESIGN AND METHODS:

Patients diagnosed with OSA at the sleep center will undergo blood pressure monitoring by measuring the blood pressure every half hour during sleep study. Patients with normal circadian BP changes are treated with CPAP as indicated. Patients with non-dipping BP pattern will be approach to join our study. The patients will receive CPAP therapy. The trial period will be 6 weeks. At the end of the trial, the patients from both treatment arms will undergo a second BP monitoring according to our above-mentioned protocol (systolic, diastolic and mean BP) to determine the circadian BP changes. Apnea-Hypopnea index will be calculated to reflect on the compliance with our therapy. Thus, patients could be divided into two study groups according to their objective compliance.

Baseline population characteristics between the placebo group and CPAP group will be noted. These include apnea-hypopnea index (AHI), medications, other co morbidities and other factors that might affect the normal circadian BP dipping pattern including factors affecting the volume status i.e. diabetes, renal failure, uncontrolled diabetes. Any new medications added during the 6 weeks trial period will be noted.

STATISTICAL ANALYSIS:

The difference in daytime and nighttime BP pattern will be noted between the treated (CPAP) and the non-compliant groups. The circadian BP variation will be recorded in both groups. Changes in the circadian BP pattern will be assessed on an intention-to-treat basis. The odds ratio, p value and confidence interval will be calculated. Correlation between the dipping/non-dipping pattern with CPAP compliance, severity of OSA and number of antihypertensive drugs will be studied as well

ELIGIBILITY:
Inclusion Criteria:

1. All patients with OSA who don't meet the above mentioned exclusion criteria

Exclusion Criteria:

1. Patients who have a normal diurnal sleep pattern (i.e. decrease of more than 30% of the systolic BP at night time)
2. Patients who are on three or more antihypertensives whose blood pressure is not controlled.
3. Patients previously treated with CPAP therapy within the past 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Obstructive sleep apnea patients age over 18 years
Sampling Method: Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2008-07; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
drop of Blood pressure at night | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Suzzane El-Sayegh, MD, Principal Investigator — Staten Island University Hospital
Locations (1):
- Heart Tower, Staten Island, New York, United States